CLINICAL TRIAL: NCT07377669
Title: A Retrospective and Prospective Study: Monocompartimental Knee Arthroplasty Combined With Anterior Cruciate Ligament Reconstruction Surgery - a Pilot Study
Acronym: MONO-LCA
Status: Enrolling by invitation | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Professor, Istituto Ortopedico Rizzoli
Other Study IDs: MONO-LCA
Record Dates: First submitted 2026-01-09; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Knee Arthritis Osteoarthritis; Cruciate Ligament Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- UKA + LCA patients: Patients who underwent simultaneous anterior cruciate ligament and monocompartimental knee replacement
  Interventions: Procedure: UKA + ACLr

INTERVENTIONS:
Procedure: UKA + ACLr — Simultaneous ACL reconstruction and Unicompartmental Knee Arthroplasty

SUMMARY:
This study aims to collect datas about patient who underwent simultaneous monocompartimental knee replacement and anterior cruciate ligament recontruction

DETAILED DESCRIPTION:
The aim is to understand if anterior cruciate ligament recontruction is mandatory in case of monocompartimental knee replacement, given the fact that anterior stability could be compromised at first in ACL (anterior cruciate ligament) deficient knees. Current datas in literature are not sufficient to establish if ACL must always be recontructed or if only in some cases

ELIGIBILITY:
Inclusion Criteria:

* monocompartimental knee arthrosis and ACL complete lesion
* High functional request
* Follow up >12 m
* Complete clinical and radiographic documentation
* Patients who accepted to partecipate to the study
* Patients who did non underwent surgical procedures in the controlateral knee

Exclusion Criteria:

* two stage surgeries (UKA and ACLr)
* patients affected by neuromuscolar disorders, or psychomotor disorders
* further knee ligamentous associated lesions
* revision surgery
* low functional request due to comorbilities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by monocompartimental knee arthosis and ACL complete lesion in the same knee who underwent simoultaneous one stage ACLr + UKA
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tegner-Lysholm score | 12 months after surgery
  The Tegner Lysholm Knee Scoring Scale is a questionnaire used to assess knee function and symptoms, particularly in the context of ligament injuries of the knee. It evaluates eight categories: pain, swelling, instability, locking, limp, stair climbing, squatting, and need for support. Each category is scored, and the total score, out of 100, reflects overall knee function. Higher scores indicate better knee function.

SECONDARY OUTCOMES:
SF-36 | 12 months after surgery
  It consists of 36 questions assessing the patient's general health, divided into eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The score ranges from a minimum of 0 to a maximum of 100 and has been validated in Italian.
Ucla | 12 months after surgery
  It is a questionnaire used to define activity levels after knee arthroplasty. It is patient-reported and provides a score ranging from 1 to 10. It has also been validated in Italian.
Return to Sport | 12 months after surgery
  Number of months elapsed before returning to sports activity (if resumed). Sports activities are classified according to Veil et al. into low-intensity, potentially low-intensity, intermediate-intensity, and high-intensity categories.
New KSS | 12 months after surgery
  A self-administered knee function and outcome assessment test. Validation in Italian is still ongoing.
Vas | 12 months after surgery
  Subjective pain assessment scale
KT-1000 | 12 months after surgery
  An objective tool for assessing anteroposterior knee laxity
ROM | 12 months after surgery
  Active and passive range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, Full Professor, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy